CLINICAL TRIAL: NCT02428049
Title: Lung Function After Curatively Intended Radiotherapy for Non-small-cell Lung Carcinoma, -Changes and Predictive Markers
Brief Title: Radiation Pneumonitis After SBRT for NSCLC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Norwegian Radium Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Janna Berg, consultant, Sykehuset i Vestfold HF
Other Study IDs: 2013/169
Record Dates: First submitted 2015-04-15; First posted 2015-04-28 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer; Radiotherapy; Lung Function Changes
MeSH Terms: conditions — Lung Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung cancer patients: Lung cancer patients in stages IA-IIIA destined to have stereotactic radiotherapy or conventional radiotherapy and chemotherapy in curative intent
  Interventions: Radiation: Stereotactic or conventional radiotherapy and chemotherapy in curative intent

INTERVENTIONS:
Radiation: Stereotactic or conventional radiotherapy and chemotherapy in curative intent

SUMMARY:
Aims:

1. Evaluate changes in lung function before and after radiotherapy for patients with NSCLC in stage I-III receiving curatively intended radiotherapy
2. To assess the predictive value of pulmonary function tests for the development of radiation pneumonitis after curative radiotherapy
3. To assess biomarkers in blood samples before, during, and after radiotherapy and correlate to the development of radiation pneumonitis
4. Investigate survival

DETAILED DESCRIPTION:
This prospective longitudinal study planned to include 70 patients with NSCLC in stages I-III who will be its own control group for changes in lung function.

It will be included patients destined to have stereotactic or concomitant chemoradiotherapy in curative intent.

Follow-up will include a physical examination by a pulmonologist, spirometry, determination of the diffusion capacity for carbon monoxide (DLCO), determination of the total lung capacity (TLC), residual volume (RV) and intrathoracic gas volume (ITGV) by body plethysmography, determination of the partial pressure of carbon dioxide (PaCO2) and oxygen (PaO2) by arterial blood gas analysis, the six-minute walking test, the Clinical COPD questionnaire, X-ray and CT scans and blood sample analysis at baseline, 4 to 6 weeks after treatment, and every 3 months thereafter until 12 months after SBRT.

Part of the project is to take blood samples. Specific blood samples will be analyzed to identify biomarkers that could predict the development of radiation-induced lung changes.

Unfortunately, fewer patients than planned were included.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Current lung cancer, not older than 8 weeks
* Received written consent
* Non small cell lung cancer
* Stage IA-IIIA
* Inoperable

Exclusion Criteria:

* Lack of consent
* Operable
* Additional cancer disease
* Small cell lung carcinoma or neuroendocrine lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung cancer patients in stages IA-IIIA
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2013-10; Primary Completion 2018-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
permanently reduced lung function | 2 years

SECONDARY OUTCOMES:
predictive value of pulmonary function tests for the development of a permanent reduction in lung function after curative radiotherapy | 2 years

OTHER OUTCOMES:
predictive value of genetic markers for permanently reduced lung function after curative radiotherapy | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Vestfold Hospital Trust, Tønsberg, Norway